CLINICAL TRIAL: NCT05950698
Title: The Assessment of Psychophysiological Markers by Analyzing the Heart Rate Variability, Blood Pressure, Anxiety and Depression, Eating Behavior, and Quality of Life Before and After Bariatric Surgery.
Brief Title: Obesity and Bariatric Surgery According to a Biopsychosocial Perspective.
Status: Recruiting | Type: Observational
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Luiz Guilherme Kraemer-Aguiar, MD, Associate Professor - Endocrinology, Department of Internal Medicine - Faculty of Medical Sciences - UERJ, Rio de Janeiro State University
Other Study IDs: 60506922.1.0000.5259
Record Dates: First submitted 2023-03-27; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Obesity; Heart Rate Variability; Anxiety Disorders; Depression; Quality of Life
Keywords: Obesity; Heart rate variability; Anxiety; Depression; Quality of Life
MeSH Terms: conditions — Obesity; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Obese patients submitted to bariatric surgery: 50 patients, both females and males, aged between 18 and 60 years, who will be submitted to bariatric surgery with Roux-en-Y reconstruction reduction gastroplasty technique.
  Patients will be evaluated for five times: before the bariatric surgery and 3-6-12-24 months after the bariatric surgery.
  Interventions: Device: Holter Faros 360° EKG (Bittium Corporation); Diagnostic Test: Beck Depression Inventory (BDI); Diagnostic Test: Hospital Anxiety and Depression Scales - HADS; Diagnostic Test: Three Factor Eating Questionnaire-R21 - TFEQ-R21; Diagnostic Test: hort-Form Health Survey-36 itens - SF-36

INTERVENTIONS:
Device: Holter Faros 360° EKG (Bittium Corporation) — Patients will lie down on the examination table, a five-lead ECG will be attached to their chest, and they should rest for 5 minutes before starting the ECG recording. ECG data will be collected for a 15-minute period Heart Rate Variability (HRV) recording will be performed between 09:00 and 12:00 in a fixed examination room to minimize environmental factors and diurnal fluctuations in autonomic nervous system functioning.
Diagnostic Test: Beck Depression Inventory (BDI) — The BDI assesses the depression severity. It will be administered before bariatric surgery at time T0 and 3-6-12-24 months after bariatric surgery (T1-T2-T3-T4).
Diagnostic Test: Hospital Anxiety and Depression Scales - HADS — The HADS assesses the anxiety and depression symptoms. It will be administered before bariatric surgery at time T0 and 3-6-12-24 months after bariatric surgery (T1-T2-T3-T4).
Diagnostic Test: Three Factor Eating Questionnaire-R21 - TFEQ-R21 — The TFEQ-R21assesses the quality of eating behavior. It will be administered before bariatric surgery at time T0 and 3-6-12-24 months after bariatric surgery (T1-T2-T3-T4).
Diagnostic Test: hort-Form Health Survey-36 itens - SF-36 — he TFEQ-R21assesses the quality of life Divided into different areas (functional capacity, general health status, pain, vitality, social aspects, emotional aspects, and mental health). It will be administered before bariatric surgery at time T0 and 3-6-12-24 months after bariatric surgery (T1-T2-T3-T4).

SUMMARY:
* The main goal of this prospective longitudinal observational study is to investigate the psychophysiological indicators by analyzing HRV, blood pressure, symptoms of anxiety and depression, eating behavior and quality of life during the follow-up of the general health status of patients with obesity undergoing the bariatric surgery by Roux-en-Y reconstruction reduction gastroplasty (GRYR) technique.
* The main question it aims to answer is: Does bariatric surgery changes the variables studied (HRV, anxiety, depression, eating behavior, quality of life)?
* Type of study: prospective longitudinal observational study
* Participant population: 50 patients, both females and males, aged between 18 and 60 years, will be submitted to bariatric surgery with Roux-en-Y reconstruction reduction gastroplasty technique.

Patients will be evaluated for five times: before the bariatric surgery and 3-6-12-24 months after the bariatric surgery.

DETAILED DESCRIPTION:
Objective: To study the psychophysiological indicators through analysis of heart rate variability (HRV), blood pressure, symptoms of anxiety and depression, eating behavior and quality of life in the follow-up of the general health status of patients with obesity submitted to the bariatric surgery by reduction gastroplasty with Roux-en-Y reconstruction (GRYR).

Methods: The investigators recruited patients of both sexes, aged 18-60 years, for whom bariatric surgery using GRYR techniques is recommended, from the Service of Integral Care for Obesity Sufferers (SAI-Ob) of the Multiuser Clinical Research Center (CePeM) of the Pedro Ernesto University Hospital (HUPE). Those taking hypoglycemic agents (biguanides, sulfonylureas, glinides, acarbose, GLP-1 analogues, SGLT-2 inhibitors, DPP-IV inhibitors, and insulin) and hyperglycemic agents (corticoids high dose thiazide diuretics, beta blockers, diazoxide and octreotide), very restrictive diets (intermittent fasting and ketogenic diet), pregnant women, history of neurological disorder, chronic pulmonary, cardiovascular, hepatic and/or renal diseases, in treatment for alcohol or drug abuse, smoking, severe psychiatric disorders (schizophrenia, bipolar disorder), vitamin B12 deficiency, iron-deficiency, anemia, neurodegenerative or cerebrovascular diseases, and those who refuse to sign the informed consent form.

Eligible patients will have a medical consultation, which will consist of a medical history and physical examination. After the consultation before and after bariatric surgery (after 3-6-12-24 months), patients will perform HRV recording for 15 minutes during a resting condition and then complete the Beck Depression Inventory (BDI), the Hospital Anxiety and Depression Scales (HADS), the Three Factor Eating Questionnaire-R21 (TFEQ-R21), and the Short-Form Health Survey- 36 items (SF-36).

The variables studied are considered to be indices of the health status of patients with obesity. The investigators hope to find changes in the examined psychophysiological measures to accurately guide the diagnostic process of the patient, in order to improve their quality of life and indirectly improve the effectiveness of bariatric surgery.

GOALS

* Study the variables that influence the general health (physical and psychological) of patients with obesity undergoing bariatric surgery;
* Improve the diagnostic process of patients with obesity by integrating psychophysiological indicators;
* Promote interdisciplinarity in the construction of personalized treatments;
* Promote research on HRV as a common factor to verify good or bad health of good or bad health;
* Additionally, the following goals are expected: a) provide training in research for undergraduate, master's and doctoral students who work on the project; b) provide the participation of resident physicians from the Comprehensive Care Service for Obesity Sufferers (SAI-Ob) of HUPE; c) present the results of the study as posters and oral presentations at scientific events; and d) publish scientific articles with the results found in indexed journals.

ELIGIBILITY:
Inclusion Criteria:

* Obese and liberated patients for the bariatric surgery.
* informed consent.
* Males and females between 18 and 60 years old .

Exclusion Criteria:

* Those taking hypoglycemic medications (biguanides, sulfonylureas, glinides, acarbose, GLP-1 analogues, SGLT-2 inhibitors, DPP-IV inhibitors, and insulin) and hyperglycemic medications (corticoids, high dose thiazide diuretics, beta blockers, diazoxide and octreotide), very restrictive diets (intermittent fasting and ketogenic diet), pregnant women, history of neurological disorder, chronic pulmonary, cardiovascular, hepatic and/or renal diseases, in treatment for alcohol or drug abuse, smoking, severe psychiatric disorders (schizophrenia, bipolar disorder), vitamin B12 deficiency, iron-deficiency, anemia, those with neurodegenerative brain disease or cerebrovascular disease, and those who refuse to sign the informed consent form.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Obese patients submitted to bariatric surgery:
  50 patients, both females and males, aged between 18 and 60 years, who will be submitted to bariatric surgery with Roux-en-Y reconstruction reduction gastroplasty technique.
  Patients will be evaluated for five times: before bariatric surgery and 3-6-12-24 months after bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-10-17 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Bariatric surgery changes measures of heart rate variability of patients | After 3-6-12-24 months after bariatric surgery
  Increased the parasympathetic activity measured through Respiratory sinus arrhythmia, High and low frequency (time domain measurements), and approximate entropy (non linear measurement) of the heart rate variability. Heart rate variability is recorded through Holter faros 360.
Bariatric surgery changes measure of anxiety | After 3-6-12-24 months after bariatric surgery
  Decreased scores on the HAD scale items assessing anxiety
Bariatric surgery changes measures of depression | After 3-6-12-24 months after bariatric surgery
  Decreased scores in the HAD scale and BDI questionnaire assessing depression
Bariatric surgery changes measures of perceived quality of life | After 3-6-12-24 months after bariatric surgery
  Increased scores in the SF-36 questionnaire which assesses the perceived quality of life

SECONDARY OUTCOMES:
Bariatric surgery changes eating behaviors | After 3-6-12-24 months after bariatric surgery
  Changes in the scores of the TFEQ-R21 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for Clinical and Experimental Research on Vascular Biology, Rio de Janeiro State University, Rio de Janeiro, Rio de Janeiro, Brazil, Brazil

IPD SHARING:
Plan to Share IPD: Undecided